CLINICAL TRIAL: NCT03081169
Title: Timing of Venous Thromboembolism Prophylaxis in Traumatic Brain Injury
Brief Title: Timing of VTE Prophylaxis in TBI
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment not started due to potential conflicting study at same institution. May renew study in the future.
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Michael Anstadt, Assistant Professor of Surgery, Loyola University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 209199
Record Dates: First submitted 2017-01-25; First posted 2017-03-16 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: TBI (Traumatic Brain Injury); VTE (Venous Thromboembolism)
MeSH Terms: conditions — Brain Injuries, Traumatic; Venous Thromboembolism | interventions — enoxaparin sodium; Enoxaparin; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early (24 hours) (Active Comparator): Patients will receive VTE prophylaxis (heparin 5000 U q 8 hrs or enoxaparin 30 mg q 12 hrs) 24 hours after injury if CT head is stable.
  Interventions: Drug: Enoxaparin Sodium 150 MG/ML Prefilled Syringe; Drug: Heparin
- Late (72 hours) (Active Comparator): Patients will receive VTE prophylaxis (heparin 5000 U q 8 hrs or enoxaparin 30 mg q 12 hrs) 72 hours after injury if CT head is stable.
  Interventions: Drug: Enoxaparin Sodium 150 MG/ML Prefilled Syringe; Drug: Heparin

INTERVENTIONS:
Drug: Enoxaparin Sodium 150 MG/ML Prefilled Syringe — The same drugs and dosages will be used in both groups, with only the timing being different
  Other Names: Lovenox
Drug: Heparin — The same drugs and dosages will be used in both groups, with only the timing being different

SUMMARY:
This study compares the efficacy and complication rates of early (24 hours) versus late (72 hours) VTE prophylaxis administration to TBI patients. Patients in both treatment groups will be monitored for development of VTE as well as complications from bleeding after commencement of VTE prophylaxis.

DETAILED DESCRIPTION:
This a randomized prospective study that compares the efficacy and complication rates of early (24 hours) versus late (72 hours) VTE prophylaxis administration to TBI patients. Patients who are identified as having an intracranial injury will be randomized to early versus late VTE prophylaxis using a 1:1 random numbers allocation. Patients in both treatment groups will be monitored for development of VTE, primarily with scheduled duplex ultrasound studies of the lower extremities. Any clinical suspicion of VTE will also be investigated with duplex ultrasound and/or CT angiogram of the chest. Patients will be monitored for development of complications from bleeding post commencement of VTE prophylaxis. Intracranial bleeding complications will be monitored by physical examination and CT scanning of the head when indicated. Patients who undergo craniotomy or craniectomy will have VTE prophylaxis started 72 hours post-surgery and will undergo CT scan of the head (to assure bleeding stabilization) prior to administration of VTE prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic brain injury
* Intracranial hemorrhage on CT scan

Exclusion Criteria:

* Under the age of 18
* Pregnant
* Die within 24 hours of admission
* Hospital stay less than 5 days
* Contraindications to enoxaparin or heparin
* Coagulopathy at 24 hours post-injury defined as INR>1.6 aPTT>2x normal, or platelet counts<50k
* Known history of VTE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2019-08-12 (Actual)

PRIMARY OUTCOMES:
VTE | Outcomes will be assessed until hospital discharge. Data will be presented at study completion with the expectation of approximately 2 years.
  Rate of venous thromboembolism (DVT or PE)

SECONDARY OUTCOMES:
Bleeding complications | Outcomes will be assessed until hospital discharge. Data will be presented at study completion with the expectation of approximately 2 years.
  Rate of expanding intracranial hemorrhage

CONTACTS AND LOCATIONS:
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No